CLINICAL TRIAL: NCT06631001
Title: The Effect of Abdominal Massage on Gastrointestinal Functions in Mechanically Ventilated Patients Receiving Enteral Nutrition in Intensive Care
Brief Title: "The Effect of Abdominal Massage on Gastrointestinal Functions in Mechanically Ventilated Patients Receiving Enteral Nutrition in Intensive Care"
Acronym: AMGF-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, YUSUF YÜCE, master student nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MersinU2024-AMGF
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Defecation Disorder; Gastrointestinal Motility Disorder; Gastrointestinal Motility and Defecation Conditions
Keywords: Abdominal massage; Gastrointestinal Motility and Defecation Conditions; Gastrointestinal Motility; Intensive care; enteral nutrition

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the intervention group receiving abdominal massage or the control group
Who Masked: Participant
Masking Description: This study is single-blind, meaning that participants are unaware of whether they are in the intervention or control group, while care providers and investigators have access to this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Massage Group (Experimental): This group consists of patients receiving abdominal massage. Abdominal massage will be administered twice a day for 15 minutes. This intervention is conducted to assess its effects on defecation frequency, gastric residual volume, and abdominal distension.
  Interventions: Other: Abdominal Massage
- Control Group (No Intervention): This group will receive standard care without abdominal massage. Measurements for bowel excretion frequency, gastric residual volume, and abdominal distension will also be conducted.

INTERVENTIONS:
Other: Abdominal Massage — Abdominal massage will be administered twice a day for 15 minutes over three days. This intervention aims to evaluate its effects on defecation frequency, gastric residual volume, and abdominal distension.
  Arms: Abdominal Massage Group

SUMMARY:
This study aims to evaluate the effects of abdominal massage on gastrointestinal functions in mechanically ventilated patients receiving enteral nutrition in intensive care units.

DETAILED DESCRIPTION:
Intensive care units (ICUs) are areas where advanced technologies and multidisciplinary care are provided together to sustain and treat critically ill patients. Patients treated in the ICU due to reasons such as inadequate gas exchange, increased respiratory workload, and inability to maintain airway patency are intubated and placed on mechanical ventilation support. ICU patients dependent on mechanical ventilators become reliant on external nutrition during the treatment process as they cannot meet their nutritional needs. In ICU patients, damage to the digestive mucosa due to stress may occur, leading to various gastrointestinal (GI) problems such as increased residual volume, diarrhea, constipation, and malnutrition. Therefore, providing accurate and adequate nutritional support is critically important in the treatment processes of ICU patients. In recent years, nutritional support has been included among therapeutic methods in ICUs. Studies have shown that appropriately timed nutritional support positively affects the clinical outcomes of patients in intensive care units. Enteral or parenteral nutrition methods can be chosen based on the patient's health status and guidelines.

For ICU patients on mechanical ventilator support, if the gastrointestinal tract is functional, enteral nutrition is frequently preferred. Enteral nutrition is the delivery of nutrients to the stomach or small intestine via a tube, catheter, or stoma. Enteral nutrition is a commonly used method for patients who cannot eat orally. It can reduce infection risk, shorten catabolic responses, the formation of gastric ulcers, and the length of hospital stay. Starting enteral nutrition within the first 48 hours for patients admitted to the ICU has been reported to shorten hospital stay and reduce mortality rates.

Although enteral nutrition has high physiological response rates, there are also risks and potential side effects. The most common GI complications encountered in patients receiving enteral nutrition are gastrointestinal complications. GI complications in enteral nutrition are influenced by many factors, including the patient's general condition, mechanical ventilation, hemodynamic parameters, and administered medications. These complications include aspiration, diarrhea, constipation, abdominal distension, and nausea/vomiting. These side effects have been observed in 62% of patients receiving this type of nutrition. Constipation is a digestive system complication that is often overlooked in ICU patients. Immobility, hypotension, the use of vasopressors and narcotics, and lack of access to appropriate conditions and facilities are among the reasons for constipation development. Constipation prolongs the duration of mechanical ventilation and increases the length of stay in ICUs. In a study evaluating enteral nutrition complications, 48.5% of the patients experienced dislodgement of their nasogastric tube, 45.5% had electrolyte imbalances, 34.5% developed hyperglycemia, 32.8% had diarrhea, 29.7% experienced constipation, 20.4% had vomiting, and 3.1% developed pulmonary aspiration.Another study found that 32% of ICU patients receiving enteral nutrition experienced increased gastric residual volume, while 46% developed gastrointestinal intolerance.

GI problems encountered in ICUs can be prevented, reduced, and patient comfort can be increased through pharmacological and non-pharmacological treatments (abdominal massage, aromatherapy, acupuncture, mobilization, etc.). A study investigating nutrition and motility issues in ICUs found that non-pharmacological methods, alongside pharmacological approaches, were also emphasized, with abdominal massage applied in 39% of cases to address motility problems. Non-pharmacological methods have various advantages over pharmacological approaches. The most important advantage of these methods is that they can be easily applied to individuals. Additionally, they offer a more cost-effective solution in terms of both patient and hospital costs.

Abdominal massage, which aims to stimulate and increase intestinal peristalsis, is performed by applying effleurage, petrissage, and vibration techniques clockwise on the abdomen for 15-20 minutes. Abdominal massage, performed by nurses, caregivers, or family members, is a safe, non-invasive method with no known side effects. This massage has been shown to be effective for those experiencing defecation issues, abdominal pain caused by gas or cramps, individuals with altered abdominal muscle tone, and those suffering from fecal incontinence or chronic constipation. Studies evaluating the effectiveness of abdominal massage in preventing GI complications in ICUs are relatively limited. A study found that abdominal massage was effective in reducing constipation and improving quality of life.A study on patients receiving enteral nutrition in neurology and neurosurgery clinics stated that abdominal massage could be used to prevent abdominal distension and increased gastric residual volume (GRV). According to a study conducted in Germany, it was reported that abdominal massage began to be used to improve GI complications in 38.8% of ICU patients.

There are studies in the literature examining the effects of abdominal massage on gastrointestinal system functions. Existing studies generally focus on the effects of abdominal massage on geriatric patient populations or evaluate it in intensive care patients with limited parameters. However, this research will specifically investigate the effects of abdominal massage on gastrointestinal system functions in patients who are mechanically ventilated and receiving enteral nutrition in the intensive care unit. The findings of this study will contribute to the adoption and standardization of abdominal massage practices by intensive care nurses in the care of this specific patient group, supported by scientific evidence. To contribute to this area in the literature, the study aims to evaluate the effects of abdominal massage on gastric residual volume, frequency of defecation, and abdominal distension in mechanically ventilated patients receiving enteral nutrition in the intensive care unit.

Three different sets of hypotheses have been established in the study. These are:

First Hypothesis Set H0: Abdominal massage applied to patients who are mechanically ventilated and receiving enteral nutrition in the intensive care unit has no effect on the frequency of defecation.

H1: Abdominal massage applied to patients who are mechanically ventilated and receiving enteral nutrition in the intensive care unit has an effect on the frequency of defecation.

Second Hypothesis Set H0: Abdominal massage applied to patients who are mechanically ventilated and receiving enteral nutrition in the intensive care unit has no effect on abdominal distension.

H1: Abdominal massage applied to patients who are mechanically ventilated and receiving enteral nutrition in the intensive care unit has an effect on abdominal distension.

Third Hypothesis Set H0: Abdominal massage applied to patients who are mechanically ventilated and receiving enteral nutrition in the intensive care unit has no effect on gastric residual volume.

H1: Abdominal massage applied to patients who are mechanically ventilated and receiving enteral nutrition in the intensive care unit has an effect on gastric residual volume.

Method* Type of Research The study is designed as a prospective, single-blind randomized controlled trial to determine the effects of abdominal massage on gastrointestinal system functions (frequency of defecation, abdominal distension, gastric residual volume) in mechanically ventilated patients receiving enteral nutrition in the intensive care unit. The research is prepared based on the 25-item checklist and flowchart included in the "Consolidated Standards of Reporting Trials (CONSORT-2017)." The study's Clinical Trials protocol registration will be done via ClinicalTrials.gov.

Location and Characteristics of the Research The research will be conducted at Mersin Toros State Hospital's general and surgical intensive care units between between January 2025 and August 2025. The internal intensive care unit at Mersin Toros State Hospital has 9 beds, while the surgical intensive care unit has 10 beds. The general intensive care unit consists of two separate rooms, with the first room containing 2 isolation rooms and a 3-bed ward system, and the second room having a 4-bed ward system separated by a wall. There are 22 nurses working in the general intensive care unit. The surgical intensive care unit is located in a single room with a 9-bed ward system, separated by walls and includes 1 isolation room. There are 24 nurses in the surgical intensive care unit, and health personnel from both units provide shared services, including a total of 8 clinical support staff, 6 cleaning staff, 1 attendant, 1 security personnel, and 1 medical secretary. The same physicians are on duty in both intensive care units, totaling 13 anesthesia specialists and 1 intensive care specialist. Both intensive care units are at level 3, and since enteral nutrition is administered cyclically, the patients are similar. The enteral nutrition planning for patients in the intensive care units will be done in cooperation with nutrition nurses and dietitians. The planned enteral nutrition will be administered and monitored by the nurses.

Randomization The listing of individuals forming the study sample will be done by an independent researcher who is not participating in the study. After obtaining consent from the relatives of patients who are willing to participate in the study and meet the criteria, the allocation of patients to the intervention or control group will be determined randomly using the website randomizer.org. Individuals included in the sampling will be listed from 1 to 70. The program will input the information that there will be two different groups of 35 individuals and that participants are numbered between 1 and 70. The program will randomly assign the two groups. The individuals listed by an independent researcher will be randomly numbered by the system (randomizer.org).

Blinding Due to the nature of the study, the researcher will not be blinded. Thus, the research will be conducted as a single-blind randomized controlled trial. Upon completion of the study, data will be entered into the computer by an independent researcher without specifying the intervention or control group, coded as groups A and B. Data analysis and the writing of the research report will be conducted by a statistician who does not know which group is which, using the codes A and B.

Data Collection Preparation of Data Collection Tools A "Data Collection Form" has been used in the data collection phase of the research. The data will be collected using a data collection form consisting of three sections: "Patient Clinical Condition Information Form," "Enteral Nutrition Monitoring Form," and "Bristol Stool Consistency Scale."

Patient Clinical Condition Information Form: This form containing patient clinical condition information has been prepared by the researcher to determine the socio-demographic characteristics of the participants after a review of the relevant literature. It includes an assessment of individual characteristics, the APACHE II (Acute Physiology and Chronic Health Evaluation) scoring system, and the Glasgow Coma Scale (GCS). Individual characteristics include age, gender, reason for admission to intensive care, chronic disease status, sedation status, intubation, and the start date of enteral nutrition.

APACHE II Scale: This scale is used for the evaluation of a patient's acute physiological and chronic health condition; it was developed to provide an objective assessment of the mortality risk, severity, and criticality of diseases in patients in the intensive care unit. The scoring range is between 12-71. As the score increases, the patient's prognosis worsens.

GCS: This will be used to assess the patient's level of consciousness. The scale assesses a patient as being in a coma if the score is between 0-3, stupor if between 3-8, confused if between 8-13, and oriented if between 13-14.

Enteral Nutrition Monitoring Form: The enteral nutrition monitoring form was created by the researcher according to the literature. This form will record the frequency of defecation, abdominal distension, GRV measurement, and the rate of intake of the nutritional solution to evaluate the effectiveness of gastrointestinal functions.

Frequency of Defecation: This is the assessment of patients' daily bowel movement status and is derived from routine patient monitoring forms in the intensive care unit.

Abdominal Distension: This is evaluated by applying pressure to the abdominal wall using the palpation method, assessing the tension of the abdominal wall during the applied pressure.

GRV Measurement: This refers to the volume of stomach contents measured by aspiration via a nasogastric tube using a syringe.

Bristol Stool Consistency Scale: Developed by a team of gastroenterologists in 1997 at the University of Bristol in England, the Bristol Stool Consistency Scale is used to assess stool form and provide information about changes in bowel habits and possible pathological conditions in the bowel. This scale is designed to classify stool into seven separate categories, reflecting an individual's bowel movements. According to the Bristol Stool Consistency Scale, Types 1 and 2 indicate constipation, Types 3 and 4 indicate normal stool, and Types 5, 6, and 7 indicate diarrhea.

Implementation of Data Collection Forms The study has two groups assigned through randomization: intervention and control. Relatives of patients meeting the research criteria will be informed about the study in the General Intensive Care and Surgical Intensive Care units at Mersin Toros State Hospital. Informed consent forms will be signed by the relatives of patients who agree to participate in the study, and the data collection forms will be implemented. Relatives in the intervention group will be informed about the procedure, and abdominal massage along with routine nursing care will be applied to the accepted patients.

Implementation Environment: The study will be conducted at the bedside in the General Intensive Care and Surgical Intensive Care Units of Mersin Toros State Hospital. To ensure patient privacy, the curtains at the bedside will be drawn. The intervention will be carried out one-on-one at the patient's bedside.

Implementation Position: In the intervention group, in addition to routine nursing care, abdominal massage will be applied while the patient's head will be elevated at an angle of 30-45° in a semi-fowler position before enteral nutrition is started. The patient should be stable during the abdominal massage, and monitoring should be conducted carefully. Routine nursing care will be applied to the control group. During enteral feeding, the head elevation will be maintained at an angle of 30-45°.

Frequency/Duration of Implementation: Based on previous studies, abdominal massage will be performed twice a day, at 15:00 and 21:00, for each patient over a total of 3 days. Each abdominal massage session will last for 15 minutes. Massage measurements will be taken afterward.

Stages of Abdominal Massage Application:

Abdominal massage consists of four fundamental movements: superficial effleurage (stroking), deep effleurage, petrissage (kneading), and vibration. Effleurage (stroking) is a technique applied with the palm or fingers over the abdominal area in both deep and superficial movements. Abdominal massage begins and ends with effleurage. During superficial effleurage, a movement is made with the palm from over the iliac bones to both sides of the pelvis and down towards the groin. Deep effleurage is applied along the ascending colon, transverse colon, and descending colon to support the movement of fecal contents through the intestines. In the petrissage technique, circular movements of the hands and fingers lift the muscle mass and compress the tissue. It is applied upwards along the ascending colon and downwards along the descending colon. It should not be repeated continuously in the same area. The vibration technique consists of vibration movements performed with the hands and fingers over the same muscle in the abdominal area. This method helps expel gas from the intestines.

Flow of the Research Process:

First Stage (Preparation Stage): A suitable environmental arrangement will be made in the General Intensive Care and Surgical Intensive Care Units of Mersin Toros State Hospital for the patients included in the intervention and control groups.

Second Stage (Application Stage): This stage will consist of four steps.

First Step: In the first step of the application, brief information about the research will be provided to the relatives of eligible patients at Mersin Toros State Hospital General Intensive Care and Surgical Intensive Care Units, and written consents will be obtained from the relatives.

Second Step: Sampling will be completed according to the inclusion, exclusion, and withdrawal criteria of the study, followed by randomization to form two randomized groups. The purpose and process of the research will be explained to the patient/relative individuals, who will then fill out the "Informed Consent Form" and the "Patient Clinical Status Information Form." Routine nursing care procedures will be applied to both groups.

Third Step: The abdominal massage procedure will be performed on the first day at 15:00. After a 30-minute break from enteral feeding, GRV measurements will be recorded using a syringe, abdominal distension measurements will be taken by palpation, and defecation counts will be recorded using the nurse observation form in the "Enteral Feeding Monitoring Form." The appearance of the stool will be evaluated by the researcher according to the "Bristol Stool Form Scale." The intervention group will receive a 15-minute abdominal massage. No intervention will be made in the control group other than routine nursing care.

Fourth Step: The abdominal massage procedure will be performed on the first day at 21:00. After a 30-minute break from enteral feeding at 20:30, GRV measurements will be recorded using a syringe, abdominal distension measurements will be taken by palpation, and defecation counts will be recorded using the nurse observation form in the "Enteral Feeding Monitoring Form." The appearance of the stool will be evaluated by the researcher according to the "Bristol Stool Form Scale." The intervention group will receive a 15-minute abdominal massage. No intervention will be made in the control group other than routine nursing care.

In the intervention group, abdominal massage will be performed for a total of 6 sessions over 3 days, twice daily, using the "Enteral Feeding Monitoring Form" and "Bristol Stool Form Scale," with measurements recorded.

In the control group, no interventions will be made other than routine nursing care throughout the 3-day process. Measurements will also be recorded using the "Enteral Feeding Monitoring Form" and "Bristol Stool Form Scale" twice a day for a total of 6 sessions. To eliminate ethical issues that may arise in the control group, abdominal massage will be performed on these patients after the data collection process of the research is completed.

Third Stage (Reporting Stage): In this stage, the statistical analysis of the data obtained from the patients will be performed, and the research report will be written.

Ethical Aspect of the Research:

The research will be conducted in accordance with the Helsinki Declaration. Written ethical approval will be obtained from the Mersin University Clinical Research Ethics Committee and written permission from the Mersin Provincial Health Directorate before data collection begins. Written permissions will also be obtained from the developers of the scales planned to be used in the research. Patient selection in the research will be based on voluntary participation. Principles of confidentiality and privacy will be observed, and patients/relatives will be informed that they can withdraw from the study at any time, after which their written consents will be obtained. Furthermore, patients will be informed that all data collected will be kept confidential and stored securely by the researcher.

Data Evaluation:

The data obtained from the research will be evaluated using appropriate statistical methods. Parametric or non-parametric tests will be used based on the normal distribution of comparative data analysis. Descriptive statistics will include counts and percentages. For normally distributed data, mean and standard deviation values will be provided, while for non-normally distributed data, minimum and maximum values along with median and 25th-75th percentiles will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients who have been intubated and are on enteral feeding for at least 5 days.
* Patients without wounds on the extremities or abdominal area.
* Patients without a history of surgical intervention or radiotherapy in the abdominal area.
* Patients without current gastrointestinal symptoms (constipation, diarrhea, vomiting, abdominal distension, or increased gastric residual volume).
* Patients without intestinal obstruction.
* Patients who have given consent through a first-degree relative.
* Patients with no contraindications for abdominal massage.
* Glasgow Coma Scale GCS > 3.
* Acute Physiology and Chronic Health Evaluation (APACHE II) score > 16

Exclusion Criteria:

* Patients receiving intermittent enteral nutrition
* Patients not on mechanical ventilation
* Patients with contraindications for abdominal massage
* Patients fed via Percutaneous Endoscopic Gastrostomy
* Patients who were intubated later
* Patients hospitalized due to postoperative reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Bowel Movements: This measure will assess the frequency of defecation during the intervention period. | Measured twice daily (morning and evening) over 3 days.
  he frequency of bowel movements will be recorded to assess gastrointestinal function, where increased frequency is considered a positive outcome.

SECONDARY OUTCOMES:
This measure will be used to determine the amount of stomach content remaining after feeding. | Measured twice daily (morning and evening) over 3 days.
  Gastric residual volume will be measured twice daily (morning and evening) for 3 consecutive days, with values ranging from 0 ml to 500 ml, where higher values indicate worse outcomes due to impaired gastric emptying

OTHER OUTCOMES:
This measure will be used to determine abdominal distension after feeding. | Measured twice daily (morning and evening) over 3 days.
  This measure will be used to determine the degree of abdominal distension during the intervention period, which may indicate gastrointestinal dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin Toros State Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) in this study

REFERENCES:
- [Background] Ikram S, Hussain E, Sarwar Zubairi AB. Nutrition in intensive care in adults review of the literature and development of evidence based feeding protocols. J Pak Med Assoc. 2016 Sep;66(9):1154-1164. PMID 27654738
- [Background] Btaiche IF, Chan LN, Pleva M, Kraft MD. Critical illness, gastrointestinal complications, and medication therapy during enteral feeding in critically ill adult patients. Nutr Clin Pract. 2010 Feb;25(1):32-49. doi: 10.1177/0884533609357565. PMID 20130156
- [Background] Kozeniecki M, Fritzshall R. Enteral Nutrition for Adults in the Hospital Setting. Nutr Clin Pract. 2015 Oct;30(5):634-51. doi: 10.1177/0884533615594012. Epub 2015 Jul 22. PMID 26203073
- [Background] Scott R, Bowling TE. Enteral tube feeding in adults. J R Coll Physicians Edinb. 2015 Mar;45(1):49-54. doi: 10.4997/JRCPE.2015.112. PMID 25874832
- [Background] Uysal N, Eser I, Akpinar H. The effect of abdominal massage on gastric residual volume: a randomized controlled trial. Gastroenterol Nurs. 2012 Mar-Apr;35(2):117-23. doi: 10.1097/SGA.0b013e31824c235a. PMID 22472671
- [Background] Hayashi M, Nishikido Y, Banno H, Michitaka T, Tachibana E, Tsukahara T. Effectiveness of registered dietitian-led management of early nutritional support in the emergency intensive care unit: a retrospective observational study. BMC Nutr. 2024 Jul 5;10(1):96. doi: 10.1186/s40795-024-00904-3. PMID 38970089
- [Background] Heyland DK, Cahill NE, Dhaliwal R, Sun X, Day AG, McClave SA. Impact of enteral feeding protocols on enteral nutrition delivery: results of a multicenter observational study. JPEN J Parenter Enteral Nutr. 2010 Nov-Dec;34(6):675-84. doi: 10.1177/0148607110364843. PMID 21097768
- [Background] Blumenstein I, Shastri YM, Stein J. Gastroenteric tube feeding: techniques, problems and solutions. World J Gastroenterol. 2014 Jul 14;20(26):8505-24. doi: 10.3748/wjg.v20.i26.8505. PMID 25024606
- [Background] Tatsumi H. Enteral tolerance in critically ill patients. J Intensive Care. 2019 May 7;7:30. doi: 10.1186/s40560-019-0378-0. eCollection 2019. PMID 31086671
- [Background] Barrett JS, Shepherd SJ, Gibson PR. Strategies to manage gastrointestinal symptoms complicating enteral feeding. JPEN J Parenter Enteral Nutr. 2009 Jan-Feb;33(1):21-6. doi: 10.1177/0148607108325073. Epub 2008 Nov 21. PMID 19028933
- [Background] Bernard AC, Magnuson B, Tsuei BJ, Swintosky M, Barnes S, Kearney PA. Defining and assessing tolerance in enteral nutrition. Nutr Clin Pract. 2004 Oct;19(5):481-6. doi: 10.1177/0115426504019005481. PMID 16215143
- [Background] Blaser AR, Starkopf J, Kirsimagi U, Deane AM. Definition, prevalence, and outcome of feeding intolerance in intensive care: a systematic review and meta-analysis. Acta Anaesthesiol Scand. 2014 Sep;58(8):914-22. doi: 10.1111/aas.12302. Epub 2014 Mar 11. PMID 24611520
- [Background] Pancorbo-Hidalgo PL, Garcia-Fernandez FP, Ramirez-Perez C. Complications associated with enteral nutrition by nasogastric tube in an internal medicine unit. J Clin Nurs. 2001 Jul;10(4):482-90. doi: 10.1046/j.1365-2702.2001.00498.x. PMID 11822496
- [Background] Mentec H, Dupont H, Bocchetti M, Cani P, Ponche F, Bleichner G. Upper digestive intolerance during enteral nutrition in critically ill patients: frequency, risk factors, and complications. Crit Care Med. 2001 Oct;29(10):1955-61. doi: 10.1097/00003246-200110000-00018. PMID 11588461
- [Background] Rohm KD, Schollhorn T, Boldt J, Wolf M, Papsdorf M, Piper SN. Nutrition support and treatment of motility disorders in critically ill patients - results of a survey on German intensive care units. Eur J Anaesthesiol. 2008 Jan;25(1):58-66. doi: 10.1017/S0265021507002657. Epub 2007 Sep 21. PMID 17888190
- [Background] Uysal N, Senel G, Karaca S, Kadiogullari N, Kocak N, Oguz G. [Symptoms seen in inpatient palliative care and impact of palliative care unit on symptom control]. Agri. 2015;27(2):104-10. doi: 10.5505/agri.2015.26214. Turkish. PMID 25944137
- [Background] Becker WC, Dorflinger L, Edmond SN, Islam L, Heapy AA, Fraenkel L. Barriers and facilitators to use of non-pharmacological treatments in chronic pain. BMC Fam Pract. 2017 Mar 20;18(1):41. doi: 10.1186/s12875-017-0608-2. PMID 28320337
- [Background] Sinclair M. The use of abdominal massage to treat chronic constipation. J Bodyw Mov Ther. 2011 Oct;15(4):436-45. doi: 10.1016/j.jbmt.2010.07.007. Epub 2010 Aug 25. PMID 21943617
- [Background] Liu Z, Sakakibara R, Odaka T, Uchiyama T, Yamamoto T, Ito T, Hattori T. Mechanism of abdominal massage for difficult defecation in a patient with myelopathy (HAM/TSP). J Neurol. 2005 Oct;252(10):1280-2. doi: 10.1007/s00415-005-0825-9. Epub 2005 May 20. No abstract available. PMID 15895308
- [Background] Preece J. Introducing abdominal massage in palliative care for the relief of constipation. Complement Ther Nurs Midwifery. 2002 May;8(2):101-5. doi: 10.1054/ctnm.2002.0610. PMID 12188155
- [Background] Birimoglu Okuyan C, Bilgili N. Effect of abdominal massage on constipation and quality of life in older adults: A randomized controlled trial. Complement Ther Med. 2019 Dec;47:102219. doi: 10.1016/j.ctim.2019.102219. Epub 2019 Oct 16. PMID 31780015
- [Background] Dehghan M, Fatehi Poor A, Mehdipoor R, Ahmadinejad M. Does abdominal massage improve gastrointestinal functions of intensive care patients with an endotracheal tube?: A randomized clinical trial. Complement Ther Clin Pract. 2018 Feb;30:122-128. doi: 10.1016/j.ctcp.2017.12.018. Epub 2017 Dec 30. PMID 29389471
- [Background] van Zanten AR. Do we need new prokinetics to reduce enteral feeding intolerance during critical illness? Crit Care. 2016 Sep 24;20(1):294. doi: 10.1186/s13054-016-1466-3. PMID 27663648
- [Background] Elpern EH, Stutz L, Peterson S, Gurka DP, Skipper A. Outcomes associated with enteral tube feedings in a medical intensive care unit. Am J Crit Care. 2004 May;13(3):221-7. PMID 15149056
- [Background] Lv G, Zhang T, Wang L, Fu X, Wang Y, Yao H, Fang H, Xia X, Yang J, Wang B, Zhang Z, Jin X, Kang Y, Cheng Y, Wu Q. Prediction of prokinetic agents in critically ill patients with feeding intolerance: a prospective observational clinical study. Front Nutr. 2023 Oct 27;10:1244517. doi: 10.3389/fnut.2023.1244517. eCollection 2023. PMID 37964927
- [Background] Ayas S, Leblebici B, Sozay S, Bayramoglu M, Niron EA. The effect of abdominal massage on bowel function in patients with spinal cord injury. Am J Phys Med Rehabil. 2006 Dec;85(12):951-5. doi: 10.1097/01.phm.0000247649.00219.c0. PMID 17117000
- [Background] Harrington KL, Haskvitz EM. Managing a patient's constipation with physical therapy. Phys Ther. 2006 Nov;86(11):1511-9. doi: 10.2522/ptj.20050347. PMID 17079751
- [Background] Wang J, Chen Y, Xue H, Chen Z, Wang Q, Zhu M, Yao J, Yuan H, Zhang X. Effect of abdominal massage on feeding intolerance in patients receiving enteral nutrition: A systematic review and meta-analysis. Nurs Open. 2023 May;10(5):2720-2733. doi: 10.1002/nop2.1537. Epub 2022 Dec 14. PMID 36517968
- [Background] Plint AC, Moher D, Morrison A, Schulz K, Altman DG, Hill C, Gaboury I. Does the CONSORT checklist improve the quality of reports of randomised controlled trials? A systematic review. Med J Aust. 2006 Sep 4;185(5):263-7. doi: 10.5694/j.1326-5377.2006.tb00557.x. PMID 16948622
- [Background] Dehghan M, Malakoutikhah A, Ghaedi Heidari F, Zakeri MA. The Effect of Abdominal Massage on Gastrointestinal Functions: a Systematic Review. Complement Ther Med. 2020 Nov;54:102553. doi: 10.1016/j.ctim.2020.102553. Epub 2020 Sep 12. PMID 33183670
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Background] Kalita M, Majewska K, Gradowska A, Karwowska K, Lawinski M. Food, mechanic and septic complications in patients enterally nutritioned in home conditions. Pol Przegl Chir. 2015 Feb 3;86(10):466-72. doi: 10.2478/pjs-2014-0083. PMID 25720105